CLINICAL TRIAL: NCT04357444
Title: Low Dose of IL-2 In Acute Respiratory DistrEss Syndrome Related to COVID-19
Acronym: LILIADE-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Iltoo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP200406; 2020-001571-32 (EudraCT Number)
Record Dates: First submitted 2020-04-10; First posted 2020-04-22 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-04

CONDITIONS: COVID 19
Keywords: COVID-19; SARS-CoV2; Acute Respiratory Distress Syndrome; Low dose of IL-2; Immunotherapy
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1: ILT101 (Experimental): ILT-101 in Subcutaneous route
  Interventions: Drug: 1: ILT101
- 2: Placebo Comparator (Placebo Comparator): Placebo in subcutaneous injections every day during 10 days
  Interventions: Drug: 2: Placebo Comparator

INTERVENTIONS:
Drug: 1: ILT101 — Subcutaneous injections, once-daily administration for 10 consecutive days.
  Arms: 1: ILT101
Drug: 2: Placebo Comparator — placebo in Subcutaneous route
  Arms: 2: Placebo Comparator

SUMMARY:
The purpose is to demonstrate the efficacy of low-dose interleukin 2 (Ld-IL2) administration in improving clinical course and oxygenation parameters in patients with SARS-CoV2-related ARDS.

DETAILED DESCRIPTION:
About 25% of hospitalized patients with SARS-CoV2 infection presented life-threatening respiratory conditions. Of these, 60% met ARDS criteria leading to death in 25% to 63% of the cases. SARS-CoV2-related ARDS is caused by a massive inflammatory cell infiltration leading to dysregulated cytokine/chemokine responses with lung immunopathological changes. To date, there is no treatment available.

Regulatory T cells (Treg) are a subpopulation of CD4+ T cells playing a crucial role in the control of immune responses, in part by preventing excessive inflammation. Depletion of Treg cells in models of lung infection or after berylium exposure exacerbated lung inflammation. In contrast, a beneficial role for Treg during early ARDS and its resolution has been observed.

Low-dose interleukin 2 (Ld-IL2) is the first therapy driving Treg-specific expansion and activation. Ld-IL2 was successfully tested in a wide range of preclinical models of inflammatory diseases, including beryllium-induced lung inflammation. Moreover, Ld-IL2 has been shown to be safe and free of serious adverse events when administered in patients with various autoimmune diseases. Importantly, in our previous work, we observed only very low concentrations of IL-2 in the blood (0.1 pg/mL [0.0-2.0]) as well as in the BAL supernatant (0.8 pg/mL [0.4-1.3]) collected from patients during the early phase of ARDS, suggesting that additional IL-2 could be beneficial for Treg expansion/activation.

Our objective is therefore to investigate the therapeutic benefit of Ld-IL2 as a Treg inducer for controlling SARS-CoV2-related ARDS.

After admission of patients to the intensive care unit at one of the recruiting centers, the eligibility criteria will be checked by the investigating physician and participation in the study will be proposed to the patient or parent/family member/trusted person. If the patient is unable to consent and there is no parent/family member/trusted person, the patient may be included in the emergency procedure.

After inclusion (J0), the patient will be randomized to one of the 2 treatment arms (low dose IL-2 or placebo).

The experimental treatment will be daily administered to the patient from D1 to D10.

The patient will be monitored daily until D28 during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years
* Laboratory (RT-PCR) confirmed infection with SARS-CoV2
* Patient is either under invasive or non-invasive mechanical ventilation (including high flow nasal oxygen therapy).
* Diagnosis of ARDS according to the Berlin definition of ARDS
* Onset of ARDS <96 hours
* Patient with French Social Security System
* A written informed consent by the designated substitute decision maker, if present. In the event of absence, the patient can be included by investigator's decision alone.

Exclusion Criteria:

* Previous history of ARDS in the last month
* Chronic respiratory diseases requiring long-term oxygen therapy and/or long-term respiratory assistance
* History of organ allograft.
* Active cancer
* Liver cirrhosis with basal Child and Pugh of C
* Pulmonary fibrosis
* Patient with end-of-life decision
* Patient not expected to survive for 24 hours
* Woman known to be pregnant, lactating or with a positive (urine or serum test) or indeterminate (serum test) pregnancy test
* Patient already enrolled in another interventional pharmacotherapy protocol on COVID-19
* Patient with known hypersensitivity to natural or recombinant Interleukin-2 or to any of the excipients
* Presence of any of the following abnormal laboratory values at screening: absolute neutrophil count (ANC) less than 1.5x109/L, AST or ALT greater than 5 x ULN, platelets <50,000 per mm3
* Use of chronic oral corticosteroids > 10 mg prednisone equivalent a day for a non-COVID-19-related condition
* Current uncontrolled autoimmune disease
* Patients with uncontrolled suspected or known active systemic bacterial or fungal infections
* Patient with severe, uncontrolled pre-existing (chronic) organ failure (myocardial, hepatic or renal)
* Vaccination with live attenuated vaccines in the month preceding the inclusion
* Patient with burns to ≥ 15% of their total body surface area
* Patient receiving extra-corporeal membrane oxygenation, high-frequency oscillatory ventilation or any form of extra-corporeal lung support
* Patient under legal protection (protection of the court, or in curatorship or guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
The PaO2/FiO2 ratio at D11 | at Day11

SECONDARY OUTCOMES:
Changes in Tregs between Baseline and Day 7 (expressed in %) | at Day0 and Day7
Number of days alive with oxygen therapy within 28 days | at Day28
Maximal oxygen rate within 28 days | at Day28
Number of days alive free of invasive or non-invasive ventilation within 28 days | At Day28
Number of days alive outside ICU within 28 days | at Day28
Number of days alive outside hospital within 28 days | at Day28
Time (in days) from randomization to death | through study completion at day 28
Mortality rate at D28 | at Day28
Difference between CRP levels at randomization and at Day 7 (or at the time of discharge if occurs before Day 7) | at Day0 and Day7 or at the time of discharge
Use of antibiotics for respiratory (proved or suspected) infection within 28 days | at Day28
Number of prone positioning sessions | throughout the follow up period at day 28
Changes in Tregs during the different visits between baseline and day 28 | at Day0, 5, 7, 11, 14 and Day28
Cytokines analysis on plasma samples at Day 0, 7 and 14 | at Day 0, 7 and 14
  To evaluate selected immune and inflammatory markers: Serum concentrations of cytokines and soluble factors related to the immune response and inflammatory processes will be evaluated and compare to baseline by multiplex immunoprofiling to analyse a larger number of molecules including at least IFNα2, IFNγ, IL-1α, IL-1β, IL-1RA, IL-2, IL-6, IL-8, IL-10, IL-17, TNFα, TNFβ, VEGF-A, TGF-beta, S-RAGE, SP-A, SP-D, Angiopoétine 1 and KGF.
Tregs numbers during induction period and throughout the follow up period at day 5, 7, 11, 14 and 28 compared to baseline before the first IL-2 injection. | at Day0, 5, 7, 11, 14 and Day28
Tregs percentages during induction period and throughout the follow up period at day 5, 7, 11, 14 and 28 compared to baseline before the first IL-2 injection. | at Day0, 5, 7, 11, 14 and Day28
Deep Immunophenotyping of Cellular components in blood samples at Day 0, 7, and 14 | at Day0, 7 and Day14
  Cellular components will be analysed by flow cytometry covering (i) most of the innate and adaptive immune cells including Tregs, T helper cell subsets including follicular helper cells, B cell subsets, NK cell subsets, (ii) the associated relevant markers of activation/function/differentiation, tissue migration, as well as (iii) unconventional lymphoid cells (NKT/MAIT, innate lymphoid cells), myeloid-derived suppressor cells, classical and non-classical monocytes and dendritic cells (mDC1/2, pDC).
T cell repertoire on Treg, after sorting from blood at Day 7 and Day 14 and compared to baseline | at Day0, 7 and Day14
T cell repertoire on Teff (CD4 and CD8) after sorting from blood at Day 7 and Day 14 and compared to baseline | at Day0, 7 and Day14
Single cells sequencing will be performed in BAL at Day 7 and Day 14 and compared to baseline. | at Day0, 7 and Day14

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel CONSTANTIN, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service Anesthésie Réanimation - Groupe Hospitalier Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Derived] Kakh M, Doroudchi M, Talepoor A. Induction of Regulatory T Cells After Virus Infection and Vaccination. Immunology. 2025 May 7. doi: 10.1111/imm.13927. Online ahead of print. PMID 40329764